CLINICAL TRIAL: NCT03097107
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Arm, 12-week Study to Evaluate the Safety and Efficacy of Saroglitazar Magnesium 1, 2 and 4 mg in Patients With Fasting Triglyceride ≥500 mg/dL and ≤1500 mg/dL
Brief Title: Evaluate the Safety and Efficacy of Saroglitazar Mg in Patients With Fasting Triglyceride ≥500 mg/dL and ≤1500 mg/dL
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Management decision to suspend the study due to recruitment issues
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SARO.15.001.05
Record Dates: First submitted 2017-03-24; First posted 2017-03-31 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Dyslipidemias
Keywords: hypertriglyceridemia; dyslipidemia; saroglitazar magnesium; lipid disorder
MeSH Terms: conditions — Dyslipidemias; Hypertriglyceridemia; Lipid Metabolism Disorders | interventions — saroglitazar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Saroglitazar magnesium 1 mg (Experimental): Saroglitazar magnesium 1 mg tablet orally once a day for 12 weeks
  Interventions: Drug: Saroglitazar Magnesium 1 mg
- Saroglitazar magnesium 2 mg (Experimental): Saroglitazar magnesium 2 mg tablet orally once a day for 12 weeks
  Interventions: Drug: Saroglitazar Magnesium 2 mg
- Saroglitazar magnesium 4 mg (Experimental): Saroglitazar magnesium 4 mg tablet orally once a day for 12 weeks
  Interventions: Drug: Saroglitazar Magnesium 4 mg
- Placebo (Placebo Comparator): Placebo tablet orally once a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saroglitazar Magnesium 1 mg — Randomly assigned patients will receive saroglitazar magnesium 1 mg orally once each morning before breakfast for 12 weeks
  Arms: Saroglitazar magnesium 1 mg
Drug: Saroglitazar Magnesium 2 mg — Randomly assigned patients will receive saroglitazar magnesium 2 mg orally once each morning before breakfast for 12 weeks
  Arms: Saroglitazar magnesium 2 mg
Drug: Saroglitazar Magnesium 4 mg — Randomly assigned patients will receive saroglitazar magnesium 4 mg orally once each morning before breakfast for 12 weeks
  Arms: Saroglitazar magnesium 4 mg
Drug: Placebo — Randomly assigned patients will receive placebo orally once each morning before breakfast for 12 weeks
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of Saroglitazar Magnesium 1, 2, and 4 mg in patients with fasting triglyceride ≥500 mg/dL and ≤1500 mg/dL.

DETAILED DESCRIPTION:
SARO.15.001.04 is a multicenter, prospective, randomized, double-blind, placebo-controlled, parallel arm, 12-week study designed to evaluate the safety and efficacy of Saroglitazar Magnesium 1, 2 and 4 mg in patients with fasting triglyceride ≥500 mg/dL and ≤1500 mg/dL.

A total 124 subjects will be enrolled in a ratio of 1:1:1:1 to receive either Saroglitazar Magnesium 1 mg, Saroglitazar Magnesium 2 mg, Saroglitazar Magnesium 4 mg, or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Adults subjects (≥18 year) of either gender.
2. Average fasting TG-C ≥500 mg/dL and ≤1500 mg/dL (from Visits 2 and 2.1).
3. Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. History of pancreatitis within 6 months of the initial screening visit (Visit 1); patients that have an episode of pancreatitis after Visit 1 but before randomization will not be randomized.
2. Patients with any history of pancreatitis may not be on GLP-1 agonists, DPP-4 inhibitors or pramlintide, with their last dose no sooner than 3 months prior to Visit 1; use of these agents by this population is prohibited throughout the duration of the trial and follow-up period. [Patients without a history of pancreatitis on these agents must be on a stable dose as of 3 months prior to Visit 1.]
3. History of >5% weight gain or weight loss or participation in weight gain/loss program in past 3 months and not in the maintenance phase as of Visit 1.
4. Diabetic (as per ADA guideline) patients with HbA1c >9.5 %.
5. Patients on prandial/rapid acting insulin, thiazolidinediones (TZDs) or glitazars in the 3 months prior to Visit 1.
6. Patients on unstable doses of basal insulin (i.e., glargine, detemir, NPH) with unstable defined as a greater than 20% fluctuation in daily dose within the past 3 months.
7. Patients on anti-obesity medications within 6 months of Visit 1 (orlistat, lorcaserin, phentermine, naltrexone/bupropion etc.).
8. Patients on drugs that may promote weight loss (i.e., anti-epileptic agents such as topiramate, zonisamide and the anti-depressant bupropion) may not be taken, unless the dose is stable for 3 months and the indication for use is not weight loss.
9. Patients on prohibited nutraceutical supplements contained in Annexure 1 that are unwilling to wash-out starting at Visit 1 (and abstain from use throughout the duration of the study, including follow-up).
10. Patients with unexplained hematuria prior to or first noted during Visit 1.
11. Patients with anemia who are undergoing repletion of deficiencies (iron, folate, B12) not in the maintenance phase as of Visit 1.
12. Patients on concomitant lipid-lowering medications and not willing to participate in Lead-in/Run-in Phase (Please refer Lead-in/Run-in Phase).
13. Patients having heart failure of NYHA class (III-IV), unstable angina, acute myocardial infarction, stroke, transient ischaemic attack, any coronary revascularisation procedure and hospitalization for acute coronary syndrome and discharge within 6 months prior to screening.
14. Patients with Left Ventricular dysfunction (Left Ventricular Ejection Fraction (LVEF) <40%, as measured through ECHO).
15. Uncontrolled hypertension (SBP >160 and/or DBP>100).
16. An uncontrolled thyroid disorder

    * Uncontrolled hyperthyroidism is defined as any history of hyperthyroidism that has either not been treated with either radioactive iodine (RAI) and/or surgery -or- that has been treated with RAI and/or surgery, but has required ongoing continuous or intermittent use of thyroid hormone synthesis inhibitors (i.e., methimazole or proplythiouracil) within 6 months of Visit 1.
    * Uncontrolled hypothyroidism is defined as initiation of thyroid hormone replacement therapy or dose adjustment of replacement therapy within 3 months of Visit 1.
17. History of GI malabsorption or history of gastric bypass, banding, or diversional bariatric surgery.
18. History of active liver disease or gall stones or hepatic dysfunction demonstrated by AST and ALT ≥2 times of upper normal limit (UNL) or bilirubin ≥1.5 times UNL at Visit 1.
19. History of myopathies or evidence of active muscle diseases demonstrated by CPK ≥5 times UNL at Visit 1.
20. History of any other concurrent serious illness or malignancy (except successfully treated basal and squamous cell carcinoma of the skin), within the past 5 years (e.g. tuberculosis, HIV).
21. Positive HIV, hepatitis A (positivity of IgM), hepatitis B, or hepatitis C at Visit 1.
22. History of excessive consumption of alcoholic beverages (consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking). For the remainder of the study, patients should agree to refrain from excessive alcohol consumption (i.e., >2 alcoholic beverages per day), to maintain their current dietary regimen, and to not alter their normal activity routines. (Note: patients should not drink alcohol for at least 24 hrs prior to any site visit).
23. History of known allergy, sensitivity or intolerance to the study drugs and their formulation ingredients.
24. Renal dysfunction demonstrated by abnormal eGFR <50 mL/min/1.73 m2.
25. History of clinically significant* systemic steroid therapy (intramuscular, intravenous, intra-articular, or oral route) within 3 months of the Visit 1 or anticipated requirement for systemic steroid therapy at Visit 1(however, topical, ophthalmic and inhaled steroids are allowed).

    * Clinically significant' (i.e., no more than 5 days of systemic steroids treatment within 3 months of Visit 1)
26. NSAID use in excess of a reasonably prescribed dose and/or use in individuals with a history of complications resulting from these agents.
27. Participation in any other clinical trial in the past 3 months in which investigational product was taken and/or a medical device was utilized. Patients that were screened but not randomized for another study must wait 30 days to participate in Visit 1.
28. Pregnancy (including a positive urine and serum pregnancy test at Visit 1), lactation or planned pregnancy/lactation during any time during the lead-in, study or follow-up periods.
29. Patients on hormonal contraception or hormone replacement therapy containing estrogen (progesterone based contraception and testosterone replacement therapy are permitted granted that dosing is stable for at least 3 months prior to Visit 1).
30. Women of childbearing potential (WOCBP) and men, UNLESS using effective contraceptive methods, such as an intra-uterine device or other mechanical contraception method with condom or diaphragm and spermicide) throughout the study. For male patients, contraception measures (condom and spermicide) must be taken during the study, either by the male participant or his female partner. (Note: Enrolled females otherwise must be surgically sterilize for at least the 6 months preceding Visit 1 or postmenopausal, defined as 12 months with no menses without an alternative medical cause).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2017-04-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change in triglyceride cholesterol levels | 12 Weeks
  Percentage change in triglyceride cholesterol levels from baseline to Week 12.

SECONDARY OUTCOMES:
Percentage change in TG-C | 8 Weeks
  Percentage change from baseline to Week 4 and 8 in TG-C
Percentage change in lipid profile. | 12 Weeks
  Percentage change from baseline to 12 in lipid profile.

CONTACTS AND LOCATIONS:
Overall Officials: Deven V Parmar, MD, Study Director — Zydus Therapeutics Inc.
Locations (33):
- United States (33):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Encompass Clinical Research, Encinitas, California
  - Integrated Research Center, San Diego, California
  - Ventura Clinical Trials, Ventura, California
  - Colorado Springs Health Partners, Colorado Springs, Colorado
  - Meridien Research - Bradenton, Bradenton, Florida
  - Meridien Research - Lakeland, Lakeland, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Meridien Research - Tampa, Tampa, Florida
  - River Birch Research Alliance LLC, Blue Ridge, Georgia
  - Drug Studies America, Marietta, Georgia
  - Herman Clinical Research, LLC, Suwanee, Georgia
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Mercury Street Medical, Butte, Montana
  - Einstein Clinical Research, Charlotte, North Carolina
  - Triad Clinical Trials LLC, Greensboro, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Ohio Clinical Research - Lyndhurst, Lyndhurst, Ohio
  - Awasty Research Network, LLC, Marion, Ohio
  - Ohio Clinical Research, LLC - Willoughby Hills, Willoughby Hills, Ohio
  - Columbia Research Group, Inc., Portland, Oregon
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Jackson Clinic, Jackson, Tennessee
  - Pioneer Research Solutions Inc., Houston, Texas
  - National Clinical Research - Richmond, Inc, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
See above.